CLINICAL TRIAL: NCT00570960
Title: Clinical, Inflammatory, and Economic Impact of Dextran 70 in Treating Spontaneous Bacterial Peritonitis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: drug product became unavilable
Sponsor: University of Virginia (Other)
Collaborators: American Association for the Study of Liver Diseases (Other)
Responsible Party: Principal Investigator, Patrick Northup, MD, Associate Professor, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13104
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Spontaneous Bacterial Peritonitis
Keywords: Peritonitis
MeSH Terms: conditions — Peritonitis | interventions — Dextrans; Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Dextran 70 (Experimental): antibiotic therapy in addition to dextran 70, 1.0 g/kg on days one, two and three
  Interventions: Drug: Dextran 70
- 2: Standard of Care Human Albumin (Active Comparator): antibiotic therapy in addition to human albumin, 1.5 g/kg on day one and 1.0 g/kg on day three
  Interventions: Biological: human albumin

INTERVENTIONS:
Drug: Dextran 70 — dextran 70, 1.0 g/kg on days one, two and three
  Arms: 1: Dextran 70
Biological: human albumin — human albumin 1.5 g/kg on day one and 1.0 g/kg on day three
  Arms: 2: Standard of Care Human Albumin

SUMMARY:
The core of the proposal is a prospective, randomized, double-blinded, controlled study which will compare the efficacy of dextran 70 versus human albumin in the treatment of cirrhotic patients with spontaneous bacterial peritonitis (SBP). Because dextran 70, which is FDA approved for plasma volume expansion, is significantly less expensive than human albumin, this study is designed and powered to determine if dextran 70 is equivalent in clinical efficacy when compared to albumin.

Specific aims for this project are to:

1. Assess the effect of plasma volume expansion with dextran 70 on disease-specific mortality at 30 days in cirrhotic patients with spontaneous bacterial peritonitis compared to plasma volume expansion with human albumin.
2. Assess the effect of dextran 70 compared to human albumin on the prevention of renal dysfunction within 30-days of diagnosis of SBP, as measured by the calculated creatinine clearance, plasma renin activity, serum aldosterone levels, levels of brain natriuretic peptide, and further development of the hepatorenal syndrome in cirrhotic patients with spontaneous bacterial peritonitis.
3. Compare the survival to liver transplantation, treatment costs, hospitalization costs, resource utilization, and quality of life of patients with spontaneous bacterial peritonitis treated with dextran 70 and human albumin in the 30 days following diagnosis.
4. Establish a comprehensive tissue bank of blood, ascites, and urine in patients with spontaneous bacterial peritonitis for future testing and translational research.
5. Establish a clinical electronic database with web-based data entry and remote analysis capabilities linking tissue bank samples and patient outcomes related to the above clinical trials.

DETAILED DESCRIPTION:
All patients admitted to the University of Virginia Health system who have clinically or pathologically defined cirrhosis, laboratory evidence consistent with spontaneous bacterial peritonitis and clinically or radiologically accessible ascites will be screened for participation in this prospective,randomized, double-blinded, controlled trial. All patients agreeing to participate will be treated with the standard of care antibiotic and supportive therapy and will be randomized to one of two treatment regimens. Treatment arm one will consist of human albumin, 1.5 g/kg intravenously administered at the time of enrollment and 1.0 g/kg administered on day three after enrollment. Treatment arm two will consist of dextran 70, 1.0 g/kg intravenously daily for three days. Under separate informed consent from the therapeutic portion of the study, all participants will be offered enrollment into the tissue repository and prospective outcomes database. Upon consent to enroll in the repository and database, serum, ascites, and urine will be collected from participating subjects for storage and future evaluation of inflammatory and pathophysiologic factors contributing to the morbidity and mortality of SBP and HRS. Prospectively collected clinical and outcomes data will be recorded into a perpetual electronic database for future comprehensive outcomes and translational studies. Participation in either the tissue repository or perpetual clinical database will not be compulsory to enroll in the therapeutic or prophylaxis trials. Similarly, subjects can choose not be enrolled in either the database or tissue repository.

Comprehensive treatment costs incurred in both treatment arms will be collected prospectively by study personnel and used to perform a formal cost-effectiveness analysis. Micro-costing algorithms will be used to derive direct treatment and hospitalization costs for the two treatment arms. After data collection is complete, along with the primary statistical analysis, a subgroup analysis will be performed to better clarify if benefit from either treatment arm is limited to high-risk patients or other specific patient sub-populations. As the proposed project is the first prospective, randomized, double-blinded investigation into two markedly different therapeutic options for treating SBP, this study will offer the unique opportunity to study them in an objective fashion.

All participants in the study will receive standard of care antibiotic therapy and supportive care for spontaneous bacterial peritonitis. Prior to screening, a paracentesis will have been performed and the resulting ascitic fluid sent to the lab for cell count and bacterial culture. Ascites culture media will be inoculated at the bedside with at least 10ml of fluid per culture container. Once the diagnosis of SBP is established, the patient will receive a complete history and physical examination, chest and abdominal radiographs, ultrasound examination of the liver including Doppler exam of the hepatic veins, arteries, and portal vein to evaluate for thrombosis, peripheral blood laboratory testing including a complete blood count with differential, standard serum chemistry and electrolytes including blood urea nitrogen (BUN) and creatinine, liver panel assay including aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), total, direct, and indirect bilirubin, prothrombin time (PT), partial thromboplastin time (PTT), international normalized ratio (INR), plasma renin activity (PRA), serum aldosterone level, and brain natriuretic peptide (BNP) level. Peripheral blood cultures will be obtained in standard fashion as per institutional protocols with inoculation of blood and body fluid samples directly into culture media at the bedside and similarly, central line blood cultures will be obtained if applicable. Complete blood cell counts, serum chemistry, and hepatic panels will be repeated at least daily for the first three days after diagnosis and at least every other week thereafter until 30 days. Levels of PRA, aldosterone, and BNP will be measured at study entry and on days two and three in the protocol, and again at day 30. Baseline quality of life will be assessed at enrollment and at 30 days. If the subject has consented to tissue banking, samples of blood, ascites, and urine will be collected and prepared for storage by study personnel. Tissue banking samples will be collected at enrollment, 3 days, and at 30 days from each participating subject.

After initial diagnostic paracentesis performed prior to enrollment, total paracentesis will be performed (if not done on the initial paracentesis). Colloid replacement after the initial paracentesis will be with the study drug.

Further therapeutic paracentesis will not be performed until after day three of the study protocol. Diuretic therapy will be continued in patients with clinical fluid control problems at the discretion of the medical team. However, diuretic use during the first three days of the protocol will be closely recorded by study personnel. All subjects will be placed on sodium-restricted diet, 2000 mg or less per day. All subjects not allergic to cephalosporins will receive intravenous cefotaxime as per a dosing regimen based upon their serum creatinine level. Patients with allergies or sensitivities to cephalosporins will receive meropenem as per a dosing regimen based upon their serum creatinine level.

If ascites or blood cultures grow specific bacterial pathogens, antibiotic therapy will be tailored to the narrowest spectrum antibiotic necessary for adequate coverage, based on in vitro organism susceptibilities. If any ascites is still present, all subjects will have a repeat diagnostic paracenteses at 48 hours after diagnosis for repeat of cell counts to assess for response to therapy. If ascites and blood cultures are negative, antibiotic coverage will be continued for a total of 5 days if clinical and laboratory resolution of the infection is verified. If subjects do not respond to initial therapy as measured by ascites PMN's not decreasing by 50% after the first 48 hours of treatment, the antibiotic regimen will be modified empirically by the primary medical team caring for the patient. Once resolution of the infection is established, after 5 days of initial therapy, all patients will be placed on ciprofloxacin, 750 mg once weekly for prophylaxis which will be continued indefinitely. If the patient is sensitive or allergic to fluoroquinolones, trimethoprim / sulfamethoxazole 160/800 mg once daily for 5 days a week will be used.

Subjects randomized to treatment with human albumin will receive a total of 1.5 g/kg of albumin at the time of enrollment and 1.0 g/kg on day three of the treatment protocol. To maintain blinding, the research pharmacy will prepare the 25% albumin solution in order to be identical in volume and color to the dextran 70 through the use of a dextrose diluent. Because of the different dosing schedules between the two treatment arms in this study, equivolume placebo doses of dextrose (5%) will be given on day two when an active treatment dose is not scheduled in the albumin arm. Dextrose will be used to avoid the sodium load and potential mild plasma volume expansion associated with saline infusion.

Subjects randomized to treatment with dextran 70 will receive it as a daily intravenous dose for the three days of the treatment protocol. A total daily dose of 1.0 g/kg will be administered. Because the hemodynamic compromise is often delayed by up to 48 hours after the diagnosis of SBP, daily dosing of dextran-70, instead of a single dose regimen, is a better pharmacokinetic treatment strategy in addressing the gradually worsening hemodynamic status involved with the progression of SBP to HRS. In normal humans, 45-60% of the infused dose of dextran-70 is recovered in the urine within 48 hours and the elimination half-life is approximately 24 hours. As stated above, in order to preserve blinding, the albumin, placebo, and dextran 70 treatment will all be equivolume and visually indistinguishable. An intravenous multivitamin additive will be used in the dextran solution in order to assure that the 6% dextran and 25% albumin solutions are of the same color. This multivitamin diluent has been used successfully for the same purpose in other blinded studies at UVAHS with no adverse events or known benefits associated from the multivitamin component.

ELIGIBILITY:
Inclusion Criteria:

* Meets all criteria for SBP as outlined below:

  * Ascites fluid analysis showing greater than or equal to 250 PMN permm3 as reported by automated or manual differential cell count
  * Lack of source of secondary peritonitis (e.g. appendicitis, acute cholecystitis)
  * Lack of a ruptured hollow viscous resulting in peritoneal soilage with multiple organisms
* Age > 18
* No antibiotic treatment within seven days prior to the diagnosis of SBP (except routine prophylaxis for SBP or initial empiric antibiotics at the time of diagnosis)
* Absence of other clinical infections
* Lack of any other systemic disease that could limit lifespan to less than 90 days
* Serum creatinine <3.0 mg/dL or calculated GFR>15 ml/min
* Serum international normalized ratio (INR)<3.0

Exclusion Criteria:

* Known hypersensitivity to a component of either of the study drugs
* Unwillingness to undergo diagnostic paracentesis
* Inability or unwillingness to give informed consent for study participation
* Shock or hemodynamic instability
* Active, clinically evident gastrointestinal bleeding, excluding heme-positive stools only
* Active congestive heart failure or inability to tolerate fluid volumes of study drugs
* Uncontrolled diabetes mellitus or hyperglycemia >400 mg/dl at screening
* Evidence for organic nephropathy, e.g. proteinuria >2+ on spot urine, hematuria>15 RBC's per HPF, abnormality on renal ultrasound
* Clinical history of severe volume depletion (i.e. severe diarrhea or brisk response to diuretics) within one week of diagnosis of SBP
* Laparotomy within the past 30 days prior to diagnosis of SBP
* Peritoneovenous shunt in place (i.e. Denver or LaVeen shunt)
* Prison inmate or resident of psychiatric facility
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick G Northup, M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospitalized cirrhosis patients with SBP between September 2007 and July 2009
Groups:
- Dextran Therapy Arm: antibiotic therapy in addition to dextran 70, 1.0 g/kg on days one, two and three
  Dextran 70 : dextran 70, 1.0 g/kg on days one, two and three
- Standard of Care Albumin Arm: antibiotic therapy in addition to human albumin, 1.5 g/kg on day one and 1.0 g/kg on day three
  human albumin : human albumin 1.5 g/kg on day one and 1.0 g/kg on day three
Period: Overall Study
Arm/Group | Dextran Therapy Arm | Standard of Care Albumin Arm
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dextran Therapy Arm | Standard of Care Albumin Arm | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (7.0) | 51.8 (12.2) | 51.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: 30 Day All Cause Mortality
Description: 30 day all cause mortality
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Dextran Therapy Arm | Standard of Care Albumin Arm
Number analyzed (Participants) | 4 | 4
participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Within 30 days of study drug administration.
Arm/Group | Dextran Therapy Arm | Standard of Care Albumin Arm
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dextran Therapy Arm (N=4) | Standard of Care Albumin Arm (N=4)
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fever (Infections and infestations) | 1 (1) | 1 (1)
Hepatic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (2)
Clostridium difficle colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Excess ascites recurrence (Hepatobiliary disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early because the manufacturer of Dextran 70 ceased all production of the study drug approximately 10 months into the study. It was felt by the principle investigator that continuation of the study was impossible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No